CLINICAL TRIAL: NCT00854659
Title: A Randomized, Double-Blind, Placebo-Controlled, Multiple-Dose Study of the Safety, Tolerability and Pharmacokinetics of ABT-102 in Healthy Subjects
Brief Title: A Safety, Tolerability and Pharmacokinetic Study of ABT-102 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Wolfram Nothaft, MD / Project Director, Abbott
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M10-613
Record Dates: First submitted 2009-03-02; First posted 2009-03-03 (Estimated); Last update posted 2010-11-02 (Estimated); Status verified 2010-09

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — ABT 102

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Active Comparator): ABT-102 Tablets, 4 mg BID
  Interventions: Drug: ABT-102
- 2 (Active Comparator): ABT-102 Tablets BID, escalating dose
  Interventions: Drug: ABT-102
- 3 (Active Comparator): ABT-102 Tablets BID, escalating dose
  Interventions: Drug: ABT-102
- 4 (Placebo Comparator): Placebo Tablets, BID
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ABT-102 — BID tablets, 7 days of treatment
  Arms: 1; 2; 3
Drug: Placebo — BID tablets, 7 days of treatment
  Arms: 4

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and pharmacokinetics of three different strengths of an investigational product dosed twice a day over 7 days in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Males and Females with a condition of general good health.
* Must be willing to participate in all study-related procedures.

Exclusion Criteria:

* History of significant sensitivity to any drug.
* Allergy to soy lecithin, soybeans, soybean oil, or other soybean derivatives.
* A requirement for medications, vitamins and/or herbal supplements during the study.
* Pregnant or breast-feeding.
* History of drug or alcohol abuse.
* Positive Hepatitis or HIV test.
* History of certain medical conditions or any uncontrolled medical illness.
* History of certain gastrointestinal surgeries that may interfere with gastrointestinal motility, PH or absorption.
* Current participation in another clinical study or receipt of investigational drug within the past 6 weeks.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2009-03; Primary Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
To determine the safety and tolerability of ABT-102 vs placebo in healthy adults. | 10 days
To determine the plasma concentrations and pharmacokinetic parameters of multiple does of ABT-102 vs. placebo in healthy adults. | 10 days

SECONDARY OUTCOMES:
Exploratory analyses of Quantitive Thermosensory Testing (Warm Detection Threshold, Cold Detection Threshold, Warm Pain Threshold) done at peripheral and oral sites, will be done for ABT-102 and placebo treated subjects. | 10 days

CONTACTS AND LOCATIONS:
Locations (1):
- Site Reference ID/Investigator# 18101, Austin, Texas, United States

REFERENCES:
- [Derived] Rowbotham MC, Nothaft W, Duan RW, Wang Y, Faltynek C, McGaraughty S, Chu KL, Svensson P. Oral and cutaneous thermosensory profile of selective TRPV1 inhibition by ABT-102 in a randomized healthy volunteer trial. Pain. 2011 May;152(5):1192-1200. doi: 10.1016/j.pain.2011.01.051. Epub 2011 Mar 4. PMID 21377273